CLINICAL TRIAL: NCT06732284
Title: Study of Sleep Inertia in Major Depressive Disorder by the Psychomotor Vigilance Task
Acronym: IN-DEP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-2/EE-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Major Depression; Sleep Inertia
Keywords: psychomotor vigilance task
MeSH Terms: conditions — Depressive Disorder, Major; Idiopathic Hypersomnia | interventions — Sleep

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with sleep inertia and major depression
  Interventions: Other: Psychomotor vigilance task; Other: Video-polysomnography; Other: Sleep and activity monitoring
- Patients with major depression without sleep inertia
  Interventions: Other: Psychomotor vigilance task; Other: Video-polysomnography; Other: Sleep and activity monitoring
- Controls without mood disorders or sleep inertia
  Interventions: Other: Psychomotor vigilance task; Other: Video-polysomnography; Other: Sleep and activity monitoring

INTERVENTIONS:
Other: Psychomotor vigilance task — Five PVT tests (before sleep at 7pm, 7am, 7:30am, 8am and 11am). The PVT is a 10-minute test designed to assess the vigilance and sustained attention by measuring reaction times (RT) to visual stimuli. During the test, participants are required to monitor the computer screen and press the response button as soon as a millisecond counter appears which will stop the counter and display the RT in milliseconds. The stimuli are randomly presented.
Other: Video-polysomnography — Performed overnight as part of routine care (11 p.m. to 7 a.m.).
Other: Sleep and activity monitoring — Actimeter and sleep diary to assess the sleep-wake patterns of the participants in their natural environments over a two-week period.

SUMMARY:
The study population comprises three groups of 30 analyzable participants: Patients with sleep inertia and Major Depressive Disorder, patients with Major Depressive Disorder but without sleep inertia, and controls without mood disorders or sleep inertia. Controls will be patients referred to the Sleep Disorders and Acupuncture Unit for polysomnography as part of the screening process for a sleep disorder. Only controls presenting an apnea-hypopnea index < 15/h, a periodic leg movements index during sleep < 15/h and a total sleep time ≥ 6 hours on the video-polysomnography will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Ability to understand, write and read French Inclusion criteria for patients with major depression
* Diagnosis of depression according to DSM-5 criteria
* Suspicion of a sleep disorder requiring polysomnographic screening
* Score for IHSS items 3 and 4

  * Score ≥ 1 for group with sleep inertia
  * Score = 0 for the group without sleep inertia Inclusion criteria for controls
* No complaints of sleep inertia (score = 0 on IHSS items 3 and 4)
* No excessive daytime sleepiness (Epworth Sleepiness Scale score ≤10),
* No depressive symptoms (Hospital Anxiety Depression Scale score < 8 on items 2, 4, 6, 8, 10, 12, 14).

Exclusion Criteria:

* The patient is participating in an interventional study
* The patient is under safeguard of justice or state guardianship
* Unweaned from the following medications for at least 5 half-lives prior to inclusion: wake-promoting or psychostimulant drugs (modafinil, methylphenidate, mazindol, amphetamine, pitolisant, solriamfetol, sodium oxybate), neuroleptics, hypnotics, antidepressants, anxiolytics, antiepileptics, budipine, dopamine agonist and antagonist antiemetics (except domperidone), opiates, gabapentin, pregabalin, benzodiazepines, Z-hypnotics (zolpidem and zopiclone), monoamine oxidase inhibitors, catechol-O-methyltransferase or sedative antihistamines.
* Patients with central nervous system diseases: Parkinson's disease, mild cognitive impairment and dementia, progressive supranuclear palsy, multisystem atrophy, Huntington's chorea, amyotrophic lateral sclerosis, epilepsy, history of head trauma with loss of consciousness.
* Patients with a malignant neoplastic disease requiring therapeutic treatment in the 12months prior to the screening visit
* Other medical or psychiatric illnesses (with the exception of depression in he depression group) which, in the investigator's opinion, could interfere with the study.
* History of suicide attempt (including failed attempt), or suicidal ideation in the past month
* Chronic alcohol consumption or drug abuse in the previous 6 months
* Sleep-wake circadian rhythm disorders and presence of sleep insufficiency according to ICSD-3 criteria
* Pregnant, parturient or breast-feeding women.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population comprises three groups of 30 analyzable participants: patients with Major Depressive Disorder and sleep inertia, patients with Major Depressive Disorder and without sleep inertia, and controls without mood disorders or sleep inertia. Controls will be patients referred to the Sleep Disorders and Acupuncture Unit for polysomnography as part of the screening process for a sleep disorder. Only controls presenting an apnea-hypopnea index < 15/h, a periodic leg movements index during sleep < 15/h and a total sleep time ≥ 6 hours on the video-polysomnography will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Level of vigilance and sustained attention before and after sleep between groups | Pre-sleep at 7pm and the wake-up measurements at 7am, 7:30am, 8am and 11am
  Change in the number of omissions in the PVT test. An omission is defined as a reaction time (RT) ≥ 500 msec.

SECONDARY OUTCOMES:
The severity of sleep inertia in patients with major depression and sleep inertia | Day 0
  Measured by Idiopathic Hypersomnia Severity Scale (IHSS). Sleep inertia will be defined as severe in the case of a score ≥ 2 for both items 3 and 4 (frequent and lasting more than 30 min), absent in the case of a score = 0 for both items 3 and 4, and mild in the other cases.
Age | Day 0
  Measured in years
Sex | Day 0
  Male/female
BMI (Body Mass Index) | Day 0
  Kg/m2
Age of onset and duration of mood disorder in both patient groups | Day 0
  Years
Total sleep time (TTS) | Day 0
  Measured by polysomnography, minutes
Sleep efficiency (SE) | Day 0
  Measured by polysomnography, percentage [(total sleep time/time spent in bed) x 100]
Sleep onset latency | Day 0
  Measured by polysomnography, minutes
Percentage in sleep stage (N1, N2, N3, SP) during the night and in the hour before waking up | Day 0
  Measured by polysomnography, percentage
Wake after sleep onset (WASO) | Day 0
  Measured by polysomnography, minutes
Microarousal index | Day 0
  Measured by polysomnography, number of microarousals /hour of sleep
Apnea-hypopnea index (AHI) | Day 0
  Measured by polysomnography, number of apneas and hypopneas /hour of sleep
Index of periodic leg movements (MPJ) | Day 0
  Measured by polysomnography, number of periodic leg movements /hour of sleep
Alertness | 7pm, 7am, 7:30am, 8am and 11am)
  Karolinska Sleepiness Scale (KSS)
Daytime sleepiness | Day 1
  Epworth Sleepiness Scale (ESS)
Depressive symptoms | Day 1
  Beck Depression Inventory (BDI-II)
Fatigue | Day 1
  Fatigue Severity Scale (FSS)
Anxiety and depression | Day 1
  Hospital Anxiety Depression Scale (HADS)
Apathy | Day 1
  Apathy Evaluation Scale
Insomnia | Day 1
  Insomnia Severity Index (ISI)
Morningness-eveningness circadian preferences | Day 1
  Horne and Ostberg Circadian Typology Questionnaire
Patient-reported state of health | Day 1
  Visual analog scale (VAS), 0 (worst health imaginable) -100 (best health imaginable)
Bedtime and wake-up times (weekdays and weekends) | Week 2
  measured via actimetry and sleep diary over a two-week period two weeks
Mean sleep duration (weekdays and weekends) | Week 2
  measured via actimetry and sleep diary over a two-week period two weeks
Sleep efficiency (weekdays and weekends) | Week 2
  measured via actimetry and sleep diary over a two-week period two weeks
Sleep latency (weekdays and weekends) | Week 2
  measured via actimetry and sleep diary over a two-week period two weeks
Wake time after sleep onset | Week 2
  measured via actimetry and sleep diary over a two-week period two weeks
Number of nighttime awakenings (weekdays and weekends) | Week 2
  Measured via actimetry and sleep diary over a two-week period
Number of naps (weekdays and weekends) | Week 2
  Measured via actimetry and sleep diary over a two-week period
Duration of naps (weekdays and weekends) | Week 2
  Measured via actimetry and sleep diary over a two-week period, minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elisa EVANGELISTA, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nimes, Nîmes, France